CLINICAL TRIAL: NCT03781219
Title: A Phase I, Single Arm, Dose Escalation Study to Evaluate Safety, Pharmacokinetics and Preliminary Efficacy of HL-085 Plus Vemurafenib in Patients With BRAF V600 Mutant Advanced Solid Tumor
Brief Title: A PhaseI Study of HL-085 Plus Vemurafenib in Solid Tumor With BRAF V600 Mutation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HL-085-102
Record Dates: First submitted 2018-03-01; First posted 2018-12-19 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Vemurafenib

STUDY DESIGN:
Intervention Model Description: If no Dose-limiting toxicity (DLT) occurs in the first three subjects in Cycle 1, the dose will be escalated to the next dose level; If a DLT occurs in one of the first three subjects, three additional subjects will be enrolled for the same dose cohort, and undergo the same procedures. Dose -escalation is performed based on the scheduled dose groups until DLT occurs in two or more subjects in a dose group which consists of 3 or 6 subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HL-085 plus Vemurafenib (Experimental): HL-085 will be administered as BID with specified dose. And the Vemurafenib will be taken as the instruction in the label ( 960 mg, BID)
  Interventions: Drug: HL-085; Drug: Vemurafenib

INTERVENTIONS:
Drug: HL-085 — HL-085 ( Capsule) is one MEK inhibitor.
Drug: Vemurafenib — Vemurafenib ( Tablet) is BRAF inhibitor,
  Other Names: ZELBORAF

SUMMARY:
This is a phase I, open-label, dose escalation study to evaluate tolerability, safety, pharmacokinetics and efficacy in patients with BRAF V600 mutant advanced solid tumor by HL-085 plus Vemurafenib treatment.

ELIGIBILITY:
Inclusion Criteria:

1. BRAF V600 mutation in solid tumor.
2. One measurable lesion as defined by RECIST 1.1 criteria for solid tumors.
3. Chemotherapy, immunotherapy or radiotherapy ≥ 4 weeks prior to starting the study treatment.
4. Surgery (except for tumor biopsy) or severe trauma ≤ 14 days prior to starting the study treatment.
5. ECOG performance status of 0-1.
6. Life expectancy ≥ 3 months.
7. Ability to take the medicine orally.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Hypersensitivity to study drug ingredients or their analogues.
2. Prior therapy with MEK-inhibitor.
3. Receiving any other anti-cancer therapy at the same time .
4. Active central nervous system (CNS) lesion.
5. Bleeding symptoms at Grade 3 within 4 weeks prior to starting study treatment.
6. ECG QTcB≥480msec in screening, or history of congenital long QT syndrome；
7. Uncontrolled concomitant diseases or infectious diseases.
8. Retinal diseases (Retinal Vein Occlusion (RVO) or Retinal pigment epithelial detachment (RPED) , et al.).
9. History of HIV,HCV,HBV infection.
10. Interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis will be excluded.
11. Serum HCG test is positive.
12. Other conditions that increase the risk of study and influence the result.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | up to 12 mouths
  Number of Treatment-Related Adverse Events as Assessed by CTCAE v4.03 will be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Tian, Ph.D, Study Director — Shanghai Kechow Pharma, Inc.
Locations (4):
- China (4):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Beijing Oncology Hospital, Beijing, Beijing Municipality
  - Henan Province Oncology Hospital, Zhengzhou, Henan
  - First Affiliated Hospital, Medicine School of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shi Y, Han X, Zhao Q, Zheng Y, Chen J, Yu X, Fang J, Liu Y, Huang D, Liu T, Shen H, Luo S, Yu H, Cao Y, Zhang X, Hu P. Tunlametinib (HL-085) plus vemurafenib in patients with advanced BRAF V600-mutant solid tumors: an open-label, single-arm, multicenter, phase I study. Exp Hematol Oncol. 2024 Jun 12;13(1):60. doi: 10.1186/s40164-024-00528-0. PMID 38867257